CLINICAL TRIAL: NCT00367562
Title: Phase IV Open Label Uncontrolled Trial of the Dual Blockade of the Renin Angiotensin System With Enalapril Plus Valsartan Combined With Oral Methylprednisolone for the Treatment of Proteinuria in IGA Nephropathy
Brief Title: Inhibition of the Renin Angiotensin System Plus Corticosteroids for the Treatment of Proteinuria in IGA Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Britanico (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEREKOWA33
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2006-11-01 (Estimated); Status verified 1996-01

CONDITIONS: IGA Nephropathy
Keywords: IGA NEPHROPATHY; STEROIDS; ENALAPRIL; VALSARTAN; PROTEINURIA; IMMUNOGLOBULIN A NEPHROPATHY (IGA NEPHROPATHY)
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria

INTERVENTIONS:
Drug: ENALAPRIL VALSARTAN METHYLPREDNISONE

SUMMARY:
TO ASSESS THE EFFICACY OF THE RENIN ANGIOTENSIN SYSTEM PLUS STEROIDS TO DECREASE THE AMOUNT OF PROTEINURIA IN IGA NEPHROPATHY

DETAILED DESCRIPTION:
Patients whose proteinuria was > 0.5 g/day were to receive enalapril plus valsartan coupled with oral 0.5 g/day of methylprednisone for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTES WITH IGA NEPHROPATHY WITH PROTEINURIA OVER 0.5 G/DAY

Exclusion Criteria:

* MALIGNANCY, RENAL FAILURE

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 1996-01; Study Completion 2005-12

PRIMARY OUTCOMES:
DAILY PROTEINURIA

SECONDARY OUTCOMES:
RENAL FUNCTION AS ASSESSED BY SERUM CREATININE

CONTACTS AND LOCATIONS:
Overall Officials: hernan trimarchi, M.D., Principal Investigator — Hospital Britanico
Locations (1):
- Hospital Britanico de Buenos Aires, Buenos Aires, Buenos Aires, Argentina

REFERENCES:
- [Background] Barratt J, Feehally J. IgA nephropathy. J Am Soc Nephrol. 2005 Jul;16(7):2088-97. doi: 10.1681/ASN.2005020134. Epub 2005 Jun 1. No abstract available. PMID 15930092
- [Background] Song JH, Lee SW, Suh JH, Kim ES, Hong SB, Kim KA, Kim MJ. The effects of dual blockade of the renin-angiotensin system on urinary protein and transforming growth factor-beta excretion in 2 groups of patients with IgA and diabetic nephropathy. Clin Nephrol. 2003 Nov;60(5):318-26. doi: 10.5414/cnp60318. PMID 14640237
- [Background] Russo D, Pisani A, Balletta MM, De Nicola L, Savino FA, Andreucci M, Minutolo R. Additive antiproteinuric effect of converting enzyme inhibitor and losartan in normotensive patients with IgA nephropathy. Am J Kidney Dis. 1999 May;33(5):851-6. doi: 10.1016/s0272-6386(99)70416-6. PMID 10213639
- [Background] Russo D, Minutolo R, Pisani A, Esposito R, Signoriello G, Andreucci M, Balletta MM. Coadministration of losartan and enalapril exerts additive antiproteinuric effect in IgA nephropathy. Am J Kidney Dis. 2001 Jul;38(1):18-25. doi: 10.1053/ajkd.2001.25176. PMID 11431176
- [Background] Appel GB, Waldman M. The IgA nephropathy treatment dilemma. Kidney Int. 2006 Jun;69(11):1939-44. doi: 10.1038/sj.ki.5000434. PMID 16641925
- [Background] Yoshikawa N, Ito H, Sakai T, Takekoshi Y, Honda M, Awazu M, Ito K, Iitaka K, Koitabashi Y, Yamaoka K, Nakagawa K, Nakamura H, Matsuyama S, Seino Y, Takeda N, Hattori S, Ninomiya M. A controlled trial of combined therapy for newly diagnosed severe childhood IgA nephropathy. The Japanese Pediatric IgA Nephropathy Treatment Study Group. J Am Soc Nephrol. 1999 Jan;10(1):101-9. doi: 10.1681/ASN.V101101. PMID 9890315
- [Background] Kobayashi Y, Hiki Y, Fujii K, Kurokawa A, Tateno S. Moderately proteinuric IgA nephropathy: prognostic prediction of individual clinical courses and steroid therapy in progressive cases. Nephron. 1989;53(3):250-6. doi: 10.1159/000185753. PMID 2797345
- [Background] Katafuchi R, Ikeda K, Mizumasa T, Tanaka H, Ando T, Yanase T, Masutani K, Kubo M, Fujimi S. Controlled, prospective trial of steroid treatment in IgA nephropathy: a limitation of low-dose prednisolone therapy. Am J Kidney Dis. 2003 May;41(5):972-83. doi: 10.1016/s0272-6386(03)00194-x. PMID 12722031
- [Background] Pozzi C, Bolasco PG, Fogazzi GB, Andrulli S, Altieri P, Ponticelli C, Locatelli F. Corticosteroids in IgA nephropathy: a randomised controlled trial. Lancet. 1999 Mar 13;353(9156):883-7. doi: 10.1016/s0140-6736(98)03563-6. PMID 10093981
- [Background] Samuels JA, Strippoli GF, Craig JC, Schena FP, Molony DA. Immunosuppressive treatments for immunoglobulin A nephropathy: a meta-analysis of randomized controlled trials. Nephrology (Carlton). 2004 Aug;9(4):177-85. doi: 10.1111/j.1440-1797.2004.00255.x. PMID 15363047
- See also: Related Info — http://www.asn-online.org